CLINICAL TRIAL: NCT05615610
Title: A Randomized Controlled Clinical Trial of Transcutaneous Electrical Nerve Stimulation on Cognitive Function and Upper Limb Motor Function in People With Chronic Stroke
Brief Title: Effects of Transcutaneous Electrical Nerve Stimulation on Cognitive Function and Upper Limb Motor Function in People With Chronic Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022_TVNS_STROKE
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Chronic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- tSCS (Experimental): The participants will be received eighteen 45-minute sessions of intervention, 3 sessions per week for 6 weeks.
  Interventions: Device: tSCS
- tVNS (Experimental): The participants will be received eighteen 45-minute sessions of intervention, 3 sessions per week for 6 weeks.
  Interventions: Device: tVNS
- Control (Placebo Comparator): The participants will be received eighteen 45-minute sessions of intervention, 3 sessions per week for 6 weeks.
  Interventions: Device: Control

INTERVENTIONS:
Device: tSCS — The participants in Group A will receive tSCS (Burst mode, 9 pulses per burst, pulse frequency = 160 Hz, burst frequency = 2 Hz) with upper limb exercises. The electrical stimulation will be generated by the neurostimulator (MH8000P; MEDIHIGHTEC MEDICAL CO., LTD., Taiwan). Two 7.5 × 12.6 cm electrodes will be attached between C6 and T5 level on each side of spinal column and with 2 cm from the spine. Intensity of TENS will be individually selected by the participants according to tolerance levels.
  Arms: tSCS
Device: tVNS — The participants in Group B will receive tVNS (pulse frequency = 25Hz, pulse duration = 0.3 ms) on the cymba conchae of left outer ear with upper limb exercises.The electrical stimulation will be generated by the neurostimulator (MH8000P; MEDIHIGHTEC MEDICAL CO., LTD., Taiwan). Intensity of tVNS will be individually selected by the participants according to tolerance levels. Previous studies showed that it was effective to improve the upper limb motor function in people with stroke and cognitive function in people with mild cognitive function.
  Arms: tVNS
Device: Control — The participants in Group C will receive placebo tSCS and tVNS with upper limb exercises, where the stimulation will be delivered by placebo-TENS device with disconnected electrical circuit.
  Arms: Control

SUMMARY:
Upper limb impairment is present in more than 85% of people with stroke, which greatly affect the quality of life, social participation, and performance of daily activities of people with stroke. Previous study also revealed that 53.4% of people after stroke experienced cognitive impairment. Different cognitive domains might be affected following stroke, such as attention, memory, language, and orientation, and the problems with memory are often prominent. Yet, there is no effective treatment for the post-stroke cognitive impairment.

Transcutaneous spinal cord stimulation (tSCS) and transcutaneous vagus nerve stimulation (tVNS) are simple and non-invasive treatment to improve upper limb motor function and cognitive function. However, no existing studies have explored on the effects of tSCS and tVNS on cognitive function in people with stroke. Therefore, the purpose of this study is to evaluate the effectiveness of transcutaneous electrical nerve stimulation (TENS) on improving upper limb function and cognitive function in people with chronic stroke.

DETAILED DESCRIPTION:
This study aims to investigate the effects of three intervention protocols in people with stroke. The participants in Group A will receive tSCS on C6 and T5 level of the spine with upper limb exercises. The participants in Group B will receive tVNS on the cymba conchae of left outer ear with upper limb exercises. The participants in Group C will receive placebo stimulation with upper limb exercises.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 50 and 80;
2. have suffered from a single stroke at least 6 months;
3. had volitional control of the non-paretic arm and at least minimal antigravity movement in the paretic shoulder;

Exclusion Criteria:

1. have cardiac pacemaker or cochlear implant;
2. have other neurological diseases;
3. are taking medication that may affect measured outcomes;
4. have skin lesions, infection, or inflammation near selected position;
5. are participating in other drug/treatment programs.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment of the Upper Extremity | Baseline (0 week)
  The Fugl-Meyer Assessment of the Upper Extremity (FMA-UE) assesses the motor control, which included the reflex, synergistic and isolated movements and coordination of the upper extremity. It is a 3-point ordinal scale with 33 items and the total score ranges from 0 to 66. In this scale, "0" represents "cannot perform", "1" represents "performs partially" and "2" represents "performs fully". The higher score indicates better motor control of the upper extremity. The FMA-UE has an excellent inter-rater reliability (ICC = 0.98) in people with stroke.
Fugl-Meyer Assessment of the Upper Extremity | Mid-intervention (3 week)
  The Fugl-Meyer Assessment of the Upper Extremity (FMA-UE) assesses the motor control, which included the reflex, synergistic and isolated movements and coordination of the upper extremity. It is a 3-point ordinal scale with 33 items and the total score ranges from 0 to 66. In this scale, "0" represents "cannot perform", "1" represents "performs partially" and "2" represents "performs fully". The higher score indicates better motor control of the upper extremity. The FMA-UE has an excellent inter-rater reliability (ICC = 0.98) in people with stroke.
Fugl-Meyer Assessment of the Upper Extremity | Post-intervention (6 week)
  The Fugl-Meyer Assessment of the Upper Extremity (FMA-UE) assesses the motor control, which included the reflex, synergistic and isolated movements and coordination of the upper extremity. It is a 3-point ordinal scale with 33 items and the total score ranges from 0 to 66. In this scale, "0" represents "cannot perform", "1" represents "performs partially" and "2" represents "performs fully". The higher score indicates better motor control of the upper extremity. The FMA-UE has an excellent inter-rater reliability (ICC = 0.98) in people with stroke.
Fugl-Meyer Assessment of the Upper Extremity | 1-month follow-up (10 week)
  The Fugl-Meyer Assessment of the Upper Extremity (FMA-UE) assesses the motor control, which included the reflex, synergistic and isolated movements and coordination of the upper extremity. It is a 3-point ordinal scale with 33 items and the total score ranges from 0 to 66. In this scale, "0" represents "cannot perform", "1" represents "performs partially" and "2" represents "performs fully". The higher score indicates better motor control of the upper extremity. The FMA-UE has an excellent inter-rater reliability (ICC = 0.98) in people with stroke.
Montreal Cognitive Assessment | Baseline (0 week)
  The Montreal Cognitive Assessment (MoCA) is a screening tool to detect cognitive impairment of an individual with a total score of 30. The MoCA assesses different cognitive domains, including executive functioning, immediate and delayed memory, visuospatial abilities, attention, working memory, language, and orientation to time and place. It can identify dementia from controls with a sensitivity of 92.3% and specificity of 91.8% with a cut-off score of 22.
Montreal Cognitive Assessment | Mid-intervention (3 week)
  The Montreal Cognitive Assessment (MoCA) is a screening tool to detect cognitive impairment of an individual with a total score of 30. The MoCA assesses different cognitive domains, including executive functioning, immediate and delayed memory, visuospatial abilities, attention, working memory, language, and orientation to time and place. It can identify dementia from controls with a sensitivity of 92.3% and specificity of 91.8% with a cut-off score of 22.
Montreal Cognitive Assessment | Post-intervention (6 week)
  The Montreal Cognitive Assessment (MoCA) is a screening tool to detect cognitive impairment of an individual with a total score of 30. The MoCA assesses different cognitive domains, including executive functioning, immediate and delayed memory, visuospatial abilities, attention, working memory, language, and orientation to time and place. It can identify dementia from controls with a sensitivity of 92.3% and specificity of 91.8% with a cut-off score of 22.
Montreal Cognitive Assessment | 1-month follow-up (10 week)
  The Montreal Cognitive Assessment (MoCA) is a screening tool to detect cognitive impairment of an individual with a total score of 30. The MoCA assesses different cognitive domains, including executive functioning, immediate and delayed memory, visuospatial abilities, attention, working memory, language, and orientation to time and place. It can identify dementia from controls with a sensitivity of 92.3% and specificity of 91.8% with a cut-off score of 22.

SECONDARY OUTCOMES:
Wolf Motor Function Test | Baseline (0 week)
  The Wolf Motor Function Test (WMFT) evaluates the motor ability of upper extremity through timed and functional tasks. It consists of 17 tasks which is rated by 6-point scale which ranges from 0 (no attempt made to use the more affected upper extremity) to 5 (movement appears to be normal). The time for completing each functional task is also recorded, with a maximum of 120 seconds allow for each task. The higher score represents the better functioning level of upper extremity, Excellent test-retest reliability (ICC = 0.92 - 0.99) has been demonstrated in people with stroke.
Wolf Motor Function Test | Mid-intervention (3 week)
  The Wolf Motor Function Test (WMFT) evaluates the motor ability of upper extremity through timed and functional tasks. It consists of 17 tasks which is rated by 6-point scale which ranges from 0 (no attempt made to use the more affected upper extremity) to 5 (movement appears to be normal). The time for completing each functional task is also recorded, with a maximum of 120 seconds allow for each task. The higher score represents the better functioning level of upper extremity, Excellent test-retest reliability (ICC = 0.92 - 0.99) has been demonstrated in people with stroke.
Wolf Motor Function Test | Post-intervention (6 week)
  The Wolf Motor Function Test (WMFT) evaluates the motor ability of upper extremity through timed and functional tasks. It consists of 17 tasks which is rated by 6-point scale which ranges from 0 (no attempt made to use the more affected upper extremity) to 5 (movement appears to be normal). The time for completing each functional task is also recorded, with a maximum of 120 seconds allow for each task. The higher score represents the better functioning level of upper extremity, Excellent test-retest reliability (ICC = 0.92 - 0.99) has been demonstrated in people with stroke.
Wolf Motor Function Test | 1-month follow-up (10 week)
  The Wolf Motor Function Test (WMFT) evaluates the motor ability of upper extremity through timed and functional tasks. It consists of 17 tasks which is rated by 6-point scale which ranges from 0 (no attempt made to use the more affected upper extremity) to 5 (movement appears to be normal). The time for completing each functional task is also recorded, with a maximum of 120 seconds allow for each task. The higher score represents the better functioning level of upper extremity, Excellent test-retest reliability (ICC = 0.92 - 0.99) has been demonstrated in people with stroke.
Muscle strength | Baseline (0 week)
  A hand-held dynamometer (Model 01165; Lafayette Instrument, Indiana, USA) will be used to measure the muscle force generated by biceps brachii and triceps brachii muscles of affected and unaffected sides. The participant will be instructed to perform isometric contraction and resistance will be applied by the examiner to avoid movement of the arm during the measurement. Two trials will be performed for each muscle group and the mean force of two trials will be recorded.
Digit Span Test | 1-month follow-up (10 week)
  The Digit Span Test (DST) consists of two parts to measure the verbal short-term memory and working memory of an individual, which are digit span forwards and digit span backwards. The participants are presented with a series of numbers. In the digit span forward (DSF), they are required to repeat the numbers in forward order. In the digit span backward (DSB), they are asked to repeat the numbers in reverse order. The length of digits in each string increases from 3 to 9 in DSF and from 2 to 8 in DSB. Two trials are presented at each length. The test is interrupted when participant failed to either trial at equal digit length. If the participants correctly recall the sequence in either first and second trial, 1 point will be scored. The total score of DSF and DSB are 16 and 14 respectively. The intra-rater reliability of DSF and DSB are 0.891 and 0.598 respectively in older adults with neurocognitive disorder.
Digit Span Test | Post-intervention (6 week)
  The Digit Span Test (DST) consists of two parts to measure the verbal short-term memory and working memory of an individual, which are digit span forwards and digit span backwards. The participants are presented with a series of numbers. In the digit span forward (DSF), they are required to repeat the numbers in forward order. In the digit span backward (DSB), they are asked to repeat the numbers in reverse order. The length of digits in each string increases from 3 to 9 in DSF and from 2 to 8 in DSB. Two trials are presented at each length. The test is interrupted when participant failed to either trial at equal digit length. If the participants correctly recall the sequence in either first and second trial, 1 point will be scored. The total score of DSF and DSB are 16 and 14 respectively. The intra-rater reliability of DSF and DSB are 0.891 and 0.598 respectively in older adults with neurocognitive disorder.
Digit Span Test | Mid-intervention (3 week)
  The Digit Span Test (DST) consists of two parts to measure the verbal short-term memory and working memory of an individual, which are digit span forwards and digit span backwards. The participants are presented with a series of numbers. In the digit span forward (DSF), they are required to repeat the numbers in forward order. In the digit span backward (DSB), they are asked to repeat the numbers in reverse order. The length of digits in each string increases from 3 to 9 in DSF and from 2 to 8 in DSB. Two trials are presented at each length. The test is interrupted when participant failed to either trial at equal digit length. If the participants correctly recall the sequence in either first and second trial, 1 point will be scored. The total score of DSF and DSB are 16 and 14 respectively. The intra-rater reliability of DSF and DSB are 0.891 and 0.598 respectively in older adults with neurocognitive disorder.
Digit Span Test | Baseline (0 week)
  The Digit Span Test (DST) consists of two parts to measure the verbal short-term memory and working memory of an individual, which are digit span forwards and digit span backwards. The participants are presented with a series of numbers. In the digit span forward (DSF), they are required to repeat the numbers in forward order. In the digit span backward (DSB), they are asked to repeat the numbers in reverse order. The length of digits in each string increases from 3 to 9 in DSF and from 2 to 8 in DSB. Two trials are presented at each length. The test is interrupted when participant failed to either trial at equal digit length. If the participants correctly recall the sequence in either first and second trial, 1 point will be scored. The total score of DSF and DSB are 16 and 14 respectively. The intra-rater reliability of DSF and DSB are 0.891 and 0.598 respectively in older adults with neurocognitive disorder.
Arm Activity Measure | 1-month follow-up (10 week)
  The Arm Activity Measure (ArmA) is a 20-item questionnaire to assess the difficulties in passive and active upper limb tasks, where section A evaluates the passive function and section B evaluates the active function. It uses a 5-point Likert scale, ranging from 0 (no difficulty) to 4 (unable to do the task). The total score of section A and B are 32 and 52 respectively [59]. The higher score in ArmA indicates more difficulties experienced in activities when using upper limb. Good internal consistency (Cronbach's alpha = 0.85 - 0.96) has been shown in people with upper limb paresis.
Arm Activity Measure | Post-intervention (6 week)
  The Arm Activity Measure (ArmA) is a 20-item questionnaire to assess the difficulties in passive and active upper limb tasks, where section A evaluates the passive function and section B evaluates the active function. It uses a 5-point Likert scale, ranging from 0 (no difficulty) to 4 (unable to do the task). The total score of section A and B are 32 and 52 respectively [59]. The higher score in ArmA indicates more difficulties experienced in activities when using upper limb. Good internal consistency (Cronbach's alpha = 0.85 - 0.96) has been shown in people with upper limb paresis.
Arm Activity Measure | Mid-intervention (3 week)
  The Arm Activity Measure (ArmA) is a 20-item questionnaire to assess the difficulties in passive and active upper limb tasks, where section A evaluates the passive function and section B evaluates the active function. It uses a 5-point Likert scale, ranging from 0 (no difficulty) to 4 (unable to do the task). The total score of section A and B are 32 and 52 respectively [59]. The higher score in ArmA indicates more difficulties experienced in activities when using upper limb. Good internal consistency (Cronbach's alpha = 0.85 - 0.96) has been shown in people with upper limb paresis.
Arm Activity Measure | Baseline (0 week)
  The Arm Activity Measure (ArmA) is a 20-item questionnaire to assess the difficulties in passive and active upper limb tasks, where section A evaluates the passive function and section B evaluates the active function. It uses a 5-point Likert scale, ranging from 0 (no difficulty) to 4 (unable to do the task). The total score of section A and B are 32 and 52 respectively [59]. The higher score in ArmA indicates more difficulties experienced in activities when using upper limb. Good internal consistency (Cronbach's alpha = 0.85 - 0.96) has been shown in people with upper limb paresis.
12-item Short-Form Survey (second version) | 1-month follow-up (10 week)
  The 12-item Short-Form Survey (second version) (SF-12v2) will be used to measure the health-related quality of life of individuals. This instrument contains eight domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, emotional role, and mental health. The total score ranges from 0 to 100, with a higher score indicating better quality of life. It has good internal consistency (Cronbach's alpha = 0.48 - 0.81) and test-retest reliability (ICC = 0.67 - 0.82) in healthy adults.
12-item Short-Form Survey (second version) | Post-intervention (6 week)
  The 12-item Short-Form Survey (second version) (SF-12v2) will be used to measure the health-related quality of life of individuals. This instrument contains eight domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, emotional role, and mental health. The total score ranges from 0 to 100, with a higher score indicating better quality of life. It has good internal consistency (Cronbach's alpha = 0.48 - 0.81) and test-retest reliability (ICC = 0.67 - 0.82) in healthy adults.
12-item Short-Form Survey (second version) | Mid-intervention (3 week)
  The 12-item Short-Form Survey (second version) (SF-12v2) will be used to measure the health-related quality of life of individuals. This instrument contains eight domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, emotional role, and mental health. The total score ranges from 0 to 100, with a higher score indicating better quality of life. It has good internal consistency (Cronbach's alpha = 0.48 - 0.81) and test-retest reliability (ICC = 0.67 - 0.82) in healthy adults.
12-item Short-Form Survey (second version) | Baseline (0 week)
  The 12-item Short-Form Survey (second version) (SF-12v2) will be used to measure the health-related quality of life of individuals. This instrument contains eight domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, emotional role, and mental health. The total score ranges from 0 to 100, with a higher score indicating better quality of life. It has good internal consistency (Cronbach's alpha = 0.48 - 0.81) and test-retest reliability (ICC = 0.67 - 0.82) in healthy adults.
Oxford Participation and Activities Questionnaire | 1-month follow-up (10 week)
  The 23-item Oxford Participation and Activities Questionnaire (Ox-PAQ) evaluates participation and activity levels based on the three domains of routine activities, social engagement, and emotional well-being. Each item is measured on a 5-point Likert scale (0 = never; 1 = rarely; 2 = sometimes; 3 = often; 4 = always). The higher scores represent greater difficulties with participation and activities. Good to excellent internal consistency (Cronbach's α = 0.81 - 0.96) and test-retest reliability (ICC = 0.83 - 0.96) have been shown for this instrument in people with motor neuron disease, multiple sclerosis, and Parkinson's disease.
Oxford Participation and Activities Questionnaire | Post-intervention (6 week)
  The 23-item Oxford Participation and Activities Questionnaire (Ox-PAQ) evaluates participation and activity levels based on the three domains of routine activities, social engagement, and emotional well-being. Each item is measured on a 5-point Likert scale (0 = never; 1 = rarely; 2 = sometimes; 3 = often; 4 = always). The higher scores represent greater difficulties with participation and activities. Good to excellent internal consistency (Cronbach's α = 0.81 - 0.96) and test-retest reliability (ICC = 0.83 - 0.96) have been shown for this instrument in people with motor neuron disease, multiple sclerosis, and Parkinson's disease.
Oxford Participation and Activities Questionnaire | Mid-intervention (3 week)
  The 23-item Oxford Participation and Activities Questionnaire (Ox-PAQ) evaluates participation and activity levels based on the three domains of routine activities, social engagement, and emotional well-being. Each item is measured on a 5-point Likert scale (0 = never; 1 = rarely; 2 = sometimes; 3 = often; 4 = always). The higher scores represent greater difficulties with participation and activities. Good to excellent internal consistency (Cronbach's α = 0.81 - 0.96) and test-retest reliability (ICC = 0.83 - 0.96) have been shown for this instrument in people with motor neuron disease, multiple sclerosis, and Parkinson's disease.
Oxford Participation and Activities Questionnaire | Baseline (0 week)
  The 23-item Oxford Participation and Activities Questionnaire (Ox-PAQ) evaluates participation and activity levels based on the three domains of routine activities, social engagement, and emotional well-being. Each item is measured on a 5-point Likert scale (0 = never; 1 = rarely; 2 = sometimes; 3 = often; 4 = always). The higher scores represent greater difficulties with participation and activities. Good to excellent internal consistency (Cronbach's α = 0.81 - 0.96) and test-retest reliability (ICC = 0.83 - 0.96) have been shown for this instrument in people with motor neuron disease, multiple sclerosis, and Parkinson's disease.
Trail Making Test | 1-month follow-up (10 week)
  Trail Making Test (TMT) can assess the attention and cognitive flexibility of individuals. The test is divided into part A and part B. In part A, the circle is numbered (i.e., 1 to 25). The subjects should draw lines in numeric order of the listed circle. In part B, the circles include both numbers (i.e., 1 to 13) and words (i.e., A to L). The subjects should draw the lines in a specific sequence between number and word (i.e., 1 to A to 2 to B etc.). A shorter time recorded in the test indicated the better performance. The test-retest reliability has been tested in people with stroke (ICC = 0.94 and 0.86 for Part A and Part B, respectively).
Trail Making Test | Post-intervention (6 week)
  Trail Making Test (TMT) can assess the attention and cognitive flexibility of individuals. The test is divided into part A and part B. In part A, the circle is numbered (i.e., 1 to 25). The subjects should draw lines in numeric order of the listed circle. In part B, the circles include both numbers (i.e., 1 to 13) and words (i.e., A to L). The subjects should draw the lines in a specific sequence between number and word (i.e., 1 to A to 2 to B etc.). A shorter time recorded in the test indicated the better performance. The test-retest reliability has been tested in people with stroke (ICC = 0.94 and 0.86 for Part A and Part B, respectively).
Trail Making Test | Mid-intervention (3 week)
  Trail Making Test (TMT) can assess the attention and cognitive flexibility of individuals. The test is divided into part A and part B. In part A, the circle is numbered (i.e., 1 to 25). The subjects should draw lines in numeric order of the listed circle. In part B, the circles include both numbers (i.e., 1 to 13) and words (i.e., A to L). The subjects should draw the lines in a specific sequence between number and word (i.e., 1 to A to 2 to B etc.). A shorter time recorded in the test indicated the better performance. The test-retest reliability has been tested in people with stroke (ICC = 0.94 and 0.86 for Part A and Part B, respectively).
Trail Making Test | Baseline (0 week)
  Trail Making Test (TMT) can assess the attention and cognitive flexibility of individuals. The test is divided into part A and part B. In part A, the circle is numbered (i.e., 1 to 25). The subjects should draw lines in numeric order of the listed circle. In part B, the circles include both numbers (i.e., 1 to 13) and words (i.e., A to L). The subjects should draw the lines in a specific sequence between number and word (i.e., 1 to A to 2 to B etc.). A shorter time recorded in the test indicated the better performance. The test-retest reliability has been tested in people with stroke (ICC = 0.94 and 0.86 for Part A and Part B, respectively).
Rivermead Behavioural Memory Test - Third edition | Mid-intervention (3 week)
  The Rivermead Behavioural Memory Test - Third edition (RBMT-3) examines the everyday memory function with 14 subtests, including the assessment for visual, verbal, recall, recognition, immediate, and delayed memory. The scaled score of each subtest and total scaled score will be computed by converting raw scores based on different age group using the conversion table of original RBMT-3. The minimum and maximum values of scaled scores for every subsets are 1 and 19, respectively. Higher scaled score indicates better memory function. The RBMT-3 has demonstrated excellent inter-rater reliability (ICC = 0.997) and intra-rater reliability (ICC = 0.924) and good internal consistency (Cronbach's alpha = 0.643 - 0.832) in people with dementia, mild cognitive impairment and healthy older adults.
Rivermead Behavioural Memory Test - Third edition | Baseline (0 week)
  The Rivermead Behavioural Memory Test - Third edition (RBMT-3) examines the everyday memory function with 14 subtests, including the assessment for visual, verbal, recall, recognition, immediate, and delayed memory. The scaled score of each subtest and total scaled score will be computed by converting raw scores based on different age group using the conversion table of original RBMT-3. The minimum and maximum values of scaled scores for every subsets are 1 and 19, respectively. Higher scaled score indicates better memory function. The RBMT-3 has demonstrated excellent inter-rater reliability (ICC = 0.997) and intra-rater reliability (ICC = 0.924) and good internal consistency (Cronbach's alpha = 0.643 - 0.832) in people with dementia, mild cognitive impairment and healthy older adults.
Rivermead Behavioural Memory Test - Third edition | Post-intervention (6 week)
  The Rivermead Behavioural Memory Test - Third edition (RBMT-3) examines the everyday memory function with 14 subtests, including the assessment for visual, verbal, recall, recognition, immediate, and delayed memory. The scaled score of each subtest and total scaled score will be computed by converting raw scores based on different age group using the conversion table of original RBMT-3. The minimum and maximum values of scaled scores for every subsets are 1 and 19, respectively. Higher scaled score indicates better memory function. The RBMT-3 has demonstrated excellent inter-rater reliability (ICC = 0.997) and intra-rater reliability (ICC = 0.924) and good internal consistency (Cronbach's alpha = 0.643 - 0.832) in people with dementia, mild cognitive impairment and healthy older adults.
Rivermead Behavioural Memory Test - Third edition | 1-month follow-up (10 week)
  The Rivermead Behavioural Memory Test - Third edition (RBMT-3) examines the everyday memory function with 14 subtests, including the assessment for visual, verbal, recall, recognition, immediate, and delayed memory. The scaled score of each subtest and total scaled score will be computed by converting raw scores based on different age group using the conversion table of original RBMT-3. The minimum and maximum values of scaled scores for every subsets are 1 and 19, respectively. Higher scaled score indicates better memory function. The RBMT-3 has demonstrated excellent inter-rater reliability (ICC = 0.997) and intra-rater reliability (ICC = 0.924) and good internal consistency (Cronbach's alpha = 0.643 - 0.832) in people with dementia, mild cognitive impairment and healthy older adults.
Muscle stiffness | 1-month follow-up (10 week)
  The muscle stiffness of biceps brachii and triceps brachii muscles will be quantified by MyotonPRO device (Myoton AS, Tallinn, Estonia). The MyotonPRO device will be placed perpendicularly to the skin surface and apply mechanical impulses on the muscles to generate damped oscillations of the underlying tissue. The biceps brachii measurements will be performed at the long head of the muscle in the middle of the arm. The triceps brachii measurements will be performed at the medial head of the muscle in the middle of the arm. Muscle stiffness will be described as newton-meter (N/m), where the higher value indicates the higher stiffness of the tissue.
Muscle stiffness | Post-intervention (6 week)
  The muscle stiffness of biceps brachii and triceps brachii muscles will be quantified by MyotonPRO device (Myoton AS, Tallinn, Estonia). The MyotonPRO device will be placed perpendicularly to the skin surface and apply mechanical impulses on the muscles to generate damped oscillations of the underlying tissue. The biceps brachii measurements will be performed at the long head of the muscle in the middle of the arm. The triceps brachii measurements will be performed at the medial head of the muscle in the middle of the arm. Muscle stiffness will be described as newton-meter (N/m), where the higher value indicates the higher stiffness of the tissue.
Muscle stiffness | Mid-intervention (3 week)
  The muscle stiffness of biceps brachii and triceps brachii muscles will be quantified by MyotonPRO device (Myoton AS, Tallinn, Estonia). The MyotonPRO device will be placed perpendicularly to the skin surface and apply mechanical impulses on the muscles to generate damped oscillations of the underlying tissue. The biceps brachii measurements will be performed at the long head of the muscle in the middle of the arm. The triceps brachii measurements will be performed at the medial head of the muscle in the middle of the arm. Muscle stiffness will be described as newton-meter (N/m), where the higher value indicates the higher stiffness of the tissue.
Muscle stiffness | Baseline (0 week)
  The muscle stiffness of biceps brachii and triceps brachii muscles will be quantified by MyotonPRO device (Myoton AS, Tallinn, Estonia). The MyotonPRO device will be placed perpendicularly to the skin surface and apply mechanical impulses on the muscles to generate damped oscillations of the underlying tissue. The biceps brachii measurements will be performed at the long head of the muscle in the middle of the arm. The triceps brachii measurements will be performed at the medial head of the muscle in the middle of the arm. Muscle stiffness will be described as newton-meter (N/m), where the higher value indicates the higher stiffness of the tissue.
Muscle strength | 1-month follow-up (10 week)
  A hand-held dynamometer (Model 01165; Lafayette Instrument, Indiana, USA) will be used to measure the muscle force generated by biceps brachii and triceps brachii muscles of affected and unaffected sides. The participant will be instructed to perform isometric contraction and resistance will be applied by the examiner to avoid movement of the arm during the measurement. Two trials will be performed for each muscle group and the mean force of two trials will be recorded.
Muscle strength | Post-intervention (6 week)
  A hand-held dynamometer (Model 01165; Lafayette Instrument, Indiana, USA) will be used to measure the muscle force generated by biceps brachii and triceps brachii muscles of affected and unaffected sides. The participant will be instructed to perform isometric contraction and resistance will be applied by the examiner to avoid movement of the arm during the measurement. Two trials will be performed for each muscle group and the mean force of two trials will be recorded.
Muscle strength | Mid-intervention (3 week)
  A hand-held dynamometer (Model 01165; Lafayette Instrument, Indiana, USA) will be used to measure the muscle force generated by biceps brachii and triceps brachii muscles of affected and unaffected sides. The participant will be instructed to perform isometric contraction and resistance will be applied by the examiner to avoid movement of the arm during the measurement. Two trials will be performed for each muscle group and the mean force of two trials will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Shamay NG, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie the results reported in a publication, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 months and ending 36 months following publication.
Access Criteria: IPD of this study will be available upon reasonable request. Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose will be able to access the IPD. IPD meta-analysis will be qualified for data sharing. A proposal that describes planned analyses should be directed to the corresponding author (shamay.ng@polyu.edu.hk).

REFERENCES:
- [Background] Nakayama H, Jorgensen HS, Raaschou HO, Olsen TS. Recovery of upper extremity function in stroke patients: the Copenhagen Stroke Study. Arch Phys Med Rehabil. 1994 Apr;75(4):394-8. doi: 10.1016/0003-9993(94)90161-9. PMID 8172497
- [Background] Langhorne P, Bernhardt J, Kwakkel G. Stroke rehabilitation. Lancet. 2011 May 14;377(9778):1693-702. doi: 10.1016/S0140-6736(11)60325-5. PMID 21571152
- [Background] Nichols-Larsen DS, Clark PC, Zeringue A, Greenspan A, Blanton S. Factors influencing stroke survivors' quality of life during subacute recovery. Stroke. 2005 Jul;36(7):1480-4. doi: 10.1161/01.STR.0000170706.13595.4f. Epub 2005 Jun 9. PMID 15947263
- [Background] Desrosiers J, Noreau L, Rochette A, Bourbonnais D, Bravo G, Bourget A. Predictors of long-term participation after stroke. Disabil Rehabil. 2006 Feb 28;28(4):221-30. doi: 10.1080/09638280500158372. PMID 16467057
- [Background] Ingwersen T, Wolf S, Birke G, Schlemm E, Bartling C, Bender G, Meyer A, Nolte A, Ottes K, Pade O, Peller M, Steinmetz J, Gerloff C, Thomalla G. Long-term recovery of upper limb motor function and self-reported health: results from a multicenter observational study 1 year after discharge from rehabilitation. Neurol Res Pract. 2021 Dec 27;3(1):66. doi: 10.1186/s42466-021-00164-7. PMID 34955097
- [Background] Barbay M, Diouf M, Roussel M, Godefroy O; GRECOGVASC study group. Systematic Review and Meta-Analysis of Prevalence in Post-Stroke Neurocognitive Disorders in Hospital-Based Studies. Dement Geriatr Cogn Disord. 2018;46(5-6):322-334. doi: 10.1159/000492920. Epub 2018 Nov 30. PMID 30504699
- [Background] Al-Qazzaz NK, Ali SH, Ahmad SA, Islam S, Mohamad K. Cognitive impairment and memory dysfunction after a stroke diagnosis: a post-stroke memory assessment. Neuropsychiatr Dis Treat. 2014 Sep 9;10:1677-91. doi: 10.2147/NDT.S67184. eCollection 2014. PMID 25228808
- [Background] Sun JH, Tan L, Yu JT. Post-stroke cognitive impairment: epidemiology, mechanisms and management. Ann Transl Med. 2014 Aug;2(8):80. doi: 10.3978/j.issn.2305-5839.2014.08.05. PMID 25333055
- [Background] Lam SC, Wong YY, Woo J. Reliability and validity of the abbreviated mental test (Hong Kong version) in residential care homes. J Am Geriatr Soc. 2010 Nov;58(11):2255-7. doi: 10.1111/j.1532-5415.2010.03129.x. No abstract available. PMID 21054326
- [Background] Scherder EJ, Bouma A. Effects of transcutaneous electrical nerve stimulation on memory and behavior in Alzheimer's disease may be stage-dependent. Biol Psychiatry. 1999 Mar 15;45(6):743-9. doi: 10.1016/s0006-3223(98)00072-9. PMID 10188004
- [Background] Scherder EJ, Bouma A, Steen LM. Effects of "isolated" transcutaneous electrical nerve stimulation on memory and affective behavior in patients with probable Alzheimer's disease. Biol Psychiatry. 1998 Mar 15;43(6):417-24. doi: 10.1016/s0006-3223(97)00208-4. PMID 9532346
- [Background] Kirshblum SC, Burns SP, Biering-Sorensen F, Donovan W, Graves DE, Jha A, Johansen M, Jones L, Krassioukov A, Mulcahey MJ, Schmidt-Read M, Waring W. International standards for neurological classification of spinal cord injury (revised 2011). J Spinal Cord Med. 2011 Nov;34(6):535-46. doi: 10.1179/204577211X13207446293695. No abstract available. PMID 22330108
- [Background] Wu D, Ma J, Zhang L, Wang S, Tan B, Jia G. Effect and Safety of Transcutaneous Auricular Vagus Nerve Stimulation on Recovery of Upper Limb Motor Function in Subacute Ischemic Stroke Patients: A Randomized Pilot Study. Neural Plast. 2020 Aug 1;2020:8841752. doi: 10.1155/2020/8841752. eCollection 2020. PMID 32802039
- [Background] Wang L, Zhang J, Guo C, He J, Zhang S, Wang Y, Zhao Y, Li L, Wang J, Hou L, Li S, Wang Y, Hao L, Zhao Y, Wu M, Fang J, Rong P. The efficacy and safety of transcutaneous auricular vagus nerve stimulation in patients with mild cognitive impairment: A double blinded randomized clinical trial. Brain Stimul. 2022 Nov-Dec;15(6):1405-1414. doi: 10.1016/j.brs.2022.09.003. Epub 2022 Sep 21. PMID 36150665
- [Background] Schleiger E, Sheikh N, Rowland T, Wong A, Read S, Finnigan S. Frontal EEG delta/alpha ratio and screening for post-stroke cognitive deficits: the power of four electrodes. Int J Psychophysiol. 2014 Oct;94(1):19-24. doi: 10.1016/j.ijpsycho.2014.06.012. Epub 2014 Jun 24. PMID 24971913
- [Background] Britton JW, Frey LC, Hopp JL, Korb P, Koubeissi MZ, Lievens WE, Pestana-Knight EM, St. Louis EK, authors. St. Louis EK, Frey LC, editors. Electroencephalography (EEG): An Introductory Text and Atlas of Normal and Abnormal Findings in Adults, Children, and Infants [Internet]. Chicago: American Epilepsy Society; 2016. Available from http://www.ncbi.nlm.nih.gov/books/NBK390354/ PMID 27748095
- [Background] Sheorajpanday RV, Nagels G, Weeren AJ, van Putten MJ, De Deyn PP. Reproducibility and clinical relevance of quantitative EEG parameters in cerebral ischemia: a basic approach. Clin Neurophysiol. 2009 May;120(5):845-55. doi: 10.1016/j.clinph.2009.02.171. Epub 2009 Apr 16. PMID 19375386
- [Background] van Putten MJ. The revised brain symmetry index. Clin Neurophysiol. 2007 Nov;118(11):2362-7. doi: 10.1016/j.clinph.2007.07.019. Epub 2007 Sep 20. PMID 17888719
- [Background] Agius Anastasi A, Falzon O, Camilleri K, Vella M, Muscat R. Brain Symmetry Index in Healthy and Stroke Patients for Assessment and Prognosis. Stroke Res Treat. 2017;2017:8276136. doi: 10.1155/2017/8276136. Epub 2017 Jan 30. PMID 28251015
- [Background] Fugl-Meyer AR, Jaasko L, Leyman I, Olsson S, Steglind S. The post-stroke hemiplegic patient. 1. a method for evaluation of physical performance. Scand J Rehabil Med. 1975;7(1):13-31. PMID 1135616
- [Background] Michaelsen SM, Rocha AS, Knabben RJ, Rodrigues LP, Fernandes CG. Translation, adaptation and inter-rater reliability of the administration manual for the Fugl-Meyer assessment. Rev Bras Fisioter. 2011 Jan-Feb;15(1):80-8. PMID 21519719
- [Background] Wolf SL, Thompson PA, Morris DM, Rose DK, Winstein CJ, Taub E, Giuliani C, Pearson SL. The EXCITE trial: attributes of the Wolf Motor Function Test in patients with subacute stroke. Neurorehabil Neural Repair. 2005 Sep;19(3):194-205. doi: 10.1177/1545968305276663. PMID 16093410
- [Background] Whitall J, Savin DN Jr, Harris-Love M, Waller SM. Psychometric properties of a modified Wolf Motor Function test for people with mild and moderate upper-extremity hemiparesis. Arch Phys Med Rehabil. 2006 May;87(5):656-60. doi: 10.1016/j.apmr.2006.02.004. PMID 16635628
- [Background] Ashford S, Slade M, Turner-Stokes L. Conceptualisation and development of the arm activity measure (ArmA) for assessment of activity in the hemiparetic arm. Disabil Rehabil. 2013 Aug;35(18):1513-8. doi: 10.3109/09638288.2012.743602. Epub 2013 Jan 7. PMID 23294435
- [Background] Fong KNK, Lee KKL, Tsang ZPY, Wan JYH, Zhang YY, Lau AFC. The clinical utility, reliability and validity of the Rivermead Behavioural Memory Test-Third Edition (RBMT-3) in Hong Kong older adults with or without cognitive impairments. Neuropsychol Rehabil. 2019 Jan;29(1):144-159. doi: 10.1080/09602011.2016.1272467. Epub 2017 Jan 4. PMID 28051902
- [Background] Leung JL, Lee GT, Lam YH, Chan RC, Wu JY. The use of the Digit Span Test in screening for cognitive impairment in acute medical inpatients. Int Psychogeriatr. 2011 Dec;23(10):1569-74. doi: 10.1017/S1041610211000792. Epub 2011 May 17. PMID 21729426
- [Background] de Paula JJ, Malloy-Diniz LF, Romano-Silva MA. Reliability of working memory assessment in neurocognitive disorders: a study of the Digit Span and Corsi Block-Tapping tasks. Braz J Psychiatry. 2016 Jul-Sep;38(3):262-3. doi: 10.1590/1516-4446-2015-1879. No abstract available. PMID 27579598
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Yeung PY, Wong LL, Chan CC, Leung JL, Yung CY. A validation study of the Hong Kong version of Montreal Cognitive Assessment (HK-MoCA) in Chinese older adults in Hong Kong. Hong Kong Med J. 2014 Dec;20(6):504-10. doi: 10.12809/hkmj144219. Epub 2014 Aug 15. PMID 25125421
- [Background] REITAN RM. The relation of the trail making test to organic brain damage. J Consult Psychol. 1955 Oct;19(5):393-4. doi: 10.1037/h0044509. No abstract available. PMID 13263471
- [Background] Morley D, Dummett S, Kelly L, Dawson J, Fitzpatrick R, Jenkinson C. Validation of the Oxford Participation and Activities Questionnaire. Patient Relat Outcome Meas. 2016 Jun 15;7:73-80. doi: 10.2147/PROM.S96822. eCollection 2016. PMID 27366108
- [Background] Jenkinson C, Kelly L, Dummett S, Morley D. The Oxford Participation and Activities Questionnaire (Ox-PAQ): development of a short form and index measure. Patient Relat Outcome Meas. 2019 Jul 29;10:227-232. doi: 10.2147/PROM.S210416. eCollection 2019. PMID 31551659
- [Background] Lam ET, Lam CL, Fong DY, Huang WW. Is the SF-12 version 2 Health Survey a valid and equivalent substitute for the SF-36 version 2 Health Survey for the Chinese? J Eval Clin Pract. 2013 Feb;19(1):200-8. doi: 10.1111/j.1365-2753.2011.01800.x. Epub 2011 Nov 29. PMID 22128754
- [Derived] Chan NH, Ng SSM. Effects of transcutaneous electrical nerve stimulation on cognitive function and upper limb motor function in people with chronic stroke: a study protocol for a randomised controlled trial. BMJ Open. 2025 Dec 14;15(12):e108243. doi: 10.1136/bmjopen-2025-108243. PMID 41397750